CLINICAL TRIAL: NCT05839470
Title: A Phase II, Prospective, Multicenter Study of Cadonilimab in Combination With FOLFOXIRI and Bevacizumab as First Line Therapy for Metastatic MSS Colorectal Cancer.
Brief Title: Cadonilimab Plus FOLFOXIRI and Bevacizumab as First Line Therapy for Metastatic MSS Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-026
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Oxaliplatin; Leucovorin; Levoleucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+ FOLFOXIRI+bevacizumab (Experimental): Cadonilimab (6mg/kg, iv, Q2W, Day1)+irinotecan* 165 mg/m² iv continue for 1.5 hours, D1; oxaliplatin 85 mg/m² iv continue for 2 hours, D1; leucovorin 400 or levoleucovorin 200 mg/m² iv continue for 2 hours, D1; 5-FU 2400 mg/m² cont. inf. 48h; repeat every 2 weeks (Q2W) + bevacizumab （5mg/kg，d 1）
  Interventions: Drug: cadonilimab; Drug: irinotecan; Drug: Oxaliplatin; Drug: leucovorin or levoleucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: cadonilimab — Cadonilimab (6mg/kg, iv, Q2W, Day1)
Drug: irinotecan — irinotecan* 165 mg/m² iv continue for 1.5 hours, D1
Drug: Oxaliplatin — oxaliplatin 85 mg/m² iv continue for 2 hours,
Drug: leucovorin or levoleucovorin — leucovorin 400 or levoleucovorin 200 mg/m² iv continue for 2 hours
Drug: 5-FU — 5-FU 2400 mg/m² cont. inf. 46h

SUMMARY:
Cadonilimab is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors.

This was a phase II study of cadonilimab in combination with bevacizumab and FOLFOXIRI as first line therapy for metastatic microsatellite stable (MSS) colorectal cancer. The goal of this clinical trial is to evaluated the efficacy and safety.

DETAILED DESCRIPTION:
Cadonilimab is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors.

This was a phase II study of cadonilimab in combination with bevacizumab and FOLFOXIRI as first line therapy in patients with metastatic microsatellite stable (MSS) colorectal cancer. The goal of this clinical trial is to evaluated the efficacy and safety.

Cadonilimab (6mg/kg, iv, Q2W, Day1)+irinotecan* 165 mg/m² iv continue for 1.5 hours, D1; oxaliplatin 85 mg/m² iv continue for 2 hours, D1; leucovorin 400 or levoleucovorin 200 mg/m² iv continue for 2 hours, D1; 5-FU 2400 mg/m² cont. inf. 48h; repeat every 2 weeks (Q2W) + bevacizumab （5mg/kg，d 1）

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic pMMR or MSS colorectal adenocarcinoma. Note: MMR or MSI status will be performed locally by an immunohistochemistry (IHC) or PCR based test for eligibility.
* Patients who are naïve to systemic treatment in metastatic setting.
* Patients with previous neoadjuvant or adjuvant chemotherapy (that may have included oxaliplatin or investigational VEGF inhibitors) are eligible if the treatment was completed > 12 months before inclusion.
* Patients with the presence of at least one lesion with measurable disease as per RECIST 1.1 guidelines. Lesions in previously irradiated areas should not be considered measurable unless they have clearly progressed since the radiotherapy.
* Patients have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Patients with MSI-H colorectal adenocarcinoma as defined per local assessment using standard of care testing
* Patients with metastatic disease amenable to be resected with potentially curative surgery
* Patients who have received any systemic treatment for metastatic disease.
* Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PDL2, anti-CTLA-4 antibodies, other checkpoint inhibitors
* Patients who had received radiation within 14 days prior to the first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-19 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to two years
  RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to two years
  RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China